CLINICAL TRIAL: NCT06683222
Title: Analysis of the Mediating Role of Myokines in the Dialogue Between Muscle and Bone Tissue in a Population of Healthy Women Aged 20-89 Years
Brief Title: Mediating Role of Myokines in the Dialogue Between Muscle and Bone Tissue in a Population of Healthy Women Aged 20-89 Years
Acronym: MyOs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AO12022/2023/VB-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Bone Density
Keywords: Myokines
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: The cohort will be a sub-group derived from the 425 healthy female volunteers who will be recruited for the MONIKA study. For the MONIKA study, we expect around 350 to be recruited at the Nîmes and Montpellier sites. Among these women recruited at the Nîmes and Montpellier sites, 280 participants will be invited to take part in the MyOs study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sub-group of 280 patients derived from the MONIKA study (Other)
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: Saliva sample; Diagnostic Test: Grip test; Other: MicroFET2® maximum isometric force test; Other: Maximum isometric knee extension bench test.; Other: The SPPB (Short Physical Performance Battery); Other: The 6-minute walking test.; Other: Segmental impedancemetry examination.; Other: Indirect calorimetry test.; Other: Fardellone's questionnaire; Other: ONAPS questionnaire; Other: Dietary intake.questionnaire

INTERVENTIONS:
Diagnostic Test: Blood sample — 36 ml of blood in 3 x 7 ml dry tubes, 1 x 5 ml EDTA tube, 1 x 5 ml heparinized tube, 1 x 5 ml anti-protease tube)
Diagnostic Test: Saliva sample — 5 ml of saliva will be taken.
Diagnostic Test: Grip test — The grip strength of the dominant arm will be measured with the participant in a standing position, with the arm close to the body and the elbow at 90◦ flexion, while the non-dominant arm will be positioned alongside the body. Three measurements will be taken for the dominant hand, and the mean value will be calculated and used for analysis. One minute is allowed between each repetition, to avoid muscle fatigue. Dynamometer quality control is ensured by regularly checking known resistance values.
Other: MicroFET2® maximum isometric force test — The microFET2 device is used to test isometric force. The microFET2 dynamometer is battery-powered and ergonomically designed to fit in the palm of the hand. The system is microprocessor-controlled to provide accurate, repeatable muscle force readings. The microFET Clinical software automatically performs calculations and validity tests, and allows graphs to be generated from the data, enabling reports of different patient tests to be compared
Other: Maximum isometric knee extension bench test. — The maximal isometric knee extension strength test on a specially-adapted strength bench consists in performing 3 maximal contractions with 1 minute's rest between each test.
Other: The SPPB (Short Physical Performance Battery) — Battery of tests comprising a balance test, a walking speed test and a chair-lift test
Other: The 6-minute walking test. — Muscular function will be determined by the 6-minute walk test to assess aerobic endurance. Participants will be asked to walk for 6 min as fast as possible on a shuttle track. The distance (m) covered in 6 min will be measured. Walking speed (m/s) will be calculated as the distance (m) covered in 6 min. A walking speed <0.8 m/s has been defined as a low value.
Other: Segmental impedancemetry examination. — Segmental impedancemetry involves measuring body composition using the body's resistance to the passage of a low-intensity electric current. This test is harmless to the body.
Other: Indirect calorimetry test. — An Indirect calorimetry is the standard method for measuring energy expenditure at rest. It is based on the principle that the human body burns nutrients using O2 and producing CO2.
Other: Fardellone's questionnaire — Completion of a questionnaires on calcium intake (Fardellone)
Other: ONAPS questionnaire — The ONAPS questionnaire contains questions on physical activity and sedentariness
Other: Dietary intake.questionnaire — The dietary intake questionnaire contains questions regarding the person's eating habits - how many meals a day, where they eat, whether they eat alone, what foods they eat/drink and whether they are following a particular diet and, if so, the reasons why.

SUMMARY:
The main hypothesis is that muscle acts on bone tissue via the secretion of myokines (myostatin, follistatin, irisin). This is based on previous results showing that muscle mass in different patient populations with very different body mass indexes (anorexic or obese patients) is significantly and independently associated with bone mineral density.

DETAILED DESCRIPTION:
Bone densitometry using X-ray absorptiometry (DXA) is the reference technique for measuring Bone Mineral Density (BMD). According to the International Osteoporosis Foundation (IOF), if a single site is to be preferred, it should be the total hip or femoral neck, using a single NHANES III reference curve. It should be stressed, however, that this curve was obtained from a North American population with anthropometric parameters, notably body mass index (BMI), that differ from those of the European population, particularly the Caucasian population. Apparently, only one reference curve has been obtained in France, from the OFELY study in 1993. Given the age of this cohort and the possibility of BMI changes over time in the Caucasian population, but even more so, the impossibility of transposing this curve onto new DXAs of different brands, new reference curves need to be developed. DMS IMAGING is therefore financing the MONIKA study, with the CHU de Nîmes as sponsor.

As part of this study, some 425 healthy female volunteers aged between 20 and 89 will be recruited from three centers (Nîmes, Montpellier, Lyon). A DXA examination at various bone sites (femur, rachis, radius and whole body) will provide up-to-date normalcy curves for BMD, but also for body composition (fat and lean mass), which are currently lacking. Access to this population could also enable us to better understand bone physiology and the links that may exist between bone tissue and muscle and fat tissue.For example, the serum concentration of leptin, a hormone secreted by adipose tissue, is associated with bone mass in non-obese women.More recent data show that skeletal muscle also has a secretory activity, characterized by the production of myokines.In humans, there are various arguments in favour of myostatin's action on bone tissue.However, clinical studies in humans are very limited.Through two clinical studies, myokine levels were assessed in two populations with very different BMIs. Female patients suffering from anorexia nervosa, for example, showed decreased myostatin levels, increased follistatin levels and comparable irisin levels, in parallel with very low BMD, compared with a population of young, non-malignant women.

In obese women with high BMD, it was also shown that myostatin and follistatin levels were high, whereas irisin levels were lower than in a control population. Furthermore, the effect of lean body mass on BMD was partially mediated by irisin. These results are still preliminary, having been obtained on a small group of subjects, and merit further investigation on a representative population scale. However, there are apparently no age-dependent reference values for these myokines.

In addition to the involvement of these myokines in the muscle-bone complex, these factors could also be involved in the muscle-fat complex, since new functions are now being attributed to them, such as lipolysis, which could affect the concentrations of certain adipokines, such as leptin, which in turn could have an impact on bone formation and resorption. The main hypothesis is that muscle acts on bone tissue via the secretion of myokines (myostatin, follistatin, irisin). This is based on previous results showing that muscle mass in different patient populations with very different BMIs (anorexic or obese patients) is significantly and independently associated with BMD.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Caucasian ethnicity (Europe, Middle East, North Africa) only as there is a difference in BMD by ethnicity.
* Person affiliated with or benefiting from a social security scheme.
* Free, informed consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Fragility fracture defined as a spontaneous or low-kinetic fracture (≤ one fall from height).
* Early menopause (< 40 years), hysterectomy (complete < 40 years), primary amenorrhea (absence of menstruation before 15 years), current amenorrhea of more than 3 months without contraceptive if the patient is less than 40 years old.
* Patients on treatments: prolonged corticosteroid therapy > 3 months or > 1 g (cumulative dose).
* Immobilization of more than 3 months, less than 12 months old.
* Hip fracture in a first-degree relative.

Patients with any of the following pathologies affecting bone, muscle or adipose tissue:

* Inflammatory bowel disease (IBD: Crohn's disease, ulcerative colitis) and untreated celiac disease.
* Renal insufficiency on dialysis or patients with nephrology follow-up.
* Known hypercalciuria.
* Osteomalacia, rickets, osteogenesis imperfecta.
* Osteopathy (Paget's disease, osteopetrosis, etc.).
* Chronic inflammatory rheumatism.
* Hemopathy, neoplasia.
* Hepatic insufficiency or chronic hepatitis.
* Endocrinopathy: diabetes, dysthyroidism, hypogonadism, hypercorticism, untreated acromegaly.
* Anorexia nervosa.
* Hyperparathyroidism (even controlled).
* History of digestive surgery (bariatric, gastrectomy, digestive resection other than appendectomy, etc.).
* History of organ transplantation.
* Chronic infectious disease (HIV, etc.).
* Weight loss of more than 10 kg within 6 months.
* Paresis, marked lameness or unloading of a limb, or prolonged immobilization of more than one month in the last 12 months.
* Patients on treatments that may affect bone mass or body composition:
* Biphosphonates (Alendronate (Fosamax® and generics), Risedronate (Actonel® and generics), Zoledronate (Aclasta® and generics).
* Teriparatide (Forsteo®).
* Denosumab (Prolia®)
* Selective estrogen receptor modulators (Clomifene, Tamoxifene, Toremifene, Raloxifene).
* Anabolic steroids.
* Strontium ranelate.
* Carbamazepine.
* Phenobarbital.
* Immunosuppressants.
* Patients on anti-epileptics.
* Patients with any of the following abnormalities in the measurement area:
* Major deformities of the wrist, hip or vertebrae.
* Compression of vertebral bodies, cementoplasty.
* Prosthesis, implant (breast, buttock, etc.), foreign body.
* Hip paraosteoarthropathy.
* Injection of radiological contrast medium, barium enema, nuclear medicine examination within 10 days.
* Intensive sport (more than 10 h/week).
* Extreme BMI (BMI < 18, BMI > 35 kg/m²).
* Loss of autonomy.
* People with neurodegenerative disorders affecting their ability to give consent.
* Pregnant, parturient or breast-feeding women.
* Participation in an interventional study involving a drug or medical device or a category 1 RIPH within 3 months prior to inclusion.

Ages: 20 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients only
Enrollment: 280 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Myostatin | Baseline
  Plasma concentration of myostatin will be measured in pg/ml by Enzyme-Linked Immuno Sorbent Assay
Follistatin | Baseline
  Plasma concentration of follistatin will be measured in pg/ml by Enzyme-Linked Immuno Sorbent Assay
Irisin | Baseline
  Plasma concentration of irisin will be measured in pg/ml by Enzyme-Linked Immuno Sorbent Assay
Bone Mineral Density | Baseline
  Bone densitometry using X-ray absorptiometry (DXA) measured in g/cm²
Lean body mass | Baseline
  Impedencemetry, measured in Kg

SECONDARY OUTCOMES:
Leptin | Baseline
  Plasma concentration of leptin will be measured in pg/ml by Enzyme-Linked Immuno Sorbent Assay
Adiponecotin | Baseline
  Plasma concentration of adiponecotin will be measured in pg/ml by Enzyme-Linked Immuno Sorbent Assay
Fat mass | Baseline
  Impedencemetry, measured in Kg
Bone mineral density: impedencemetry | Baseline
  Bone densitometry will be measured by impedencemetry in g/cm²
Grip test | Baseline
  Measured by a digital dynamometer (MicroFET2)
Isometric force | Baseline
  bench test
Walking test | Baseline
  Participants will be asked to walk for 6 min as fast as possible on a shuttle track. The distance (m) covered in 6 min will be measured. Walking speed (m/s) will be calculated as the distance (m) covered in 6 min. A walking speed <0.8 m/s has been defined as a low value
Short Physical Performance Battery : Balance test | Baseline
  The person's ability to stand for 10 sec with feet in 3 different positions (together side-by-side, semi-tandem, and tandem) is tested and scored as follows :
  1. Side-by-side stance scored from 0-1
  2. Semi-tandem stance scored from 0-1
  3. Tandem stance scored from 0-2
Short Physical Performance Battery : Walking speed test | Baseline
  Two timed trials of a 3-meter or 4-meter walk (fastest recorded in seconds)
Short Physical Performance Battery : Chair lift test | Baseline
  The time taken to raise a chair 5 times is recorded in seconds.
Plasma concentration of osteocalcin, a bone remodelling marker. | Baseline
  Measured in ng/ml
Plasma concentration of serum cross-linked C-telopeptide of type I collagen (CTX), a bone remodelling marker. | Baseline
  Measured in pmol/l
Calcium intake | Baseline
  Calcium intake (mg/day) will be measured using the Fardellone Dietary intake questionnaire (protein (gr), carbohydrate (gr), fat (gr)) will be assessed using the dietary habits questionnaire.
Level of physical activity | Baseline
  Level of physical activity (hours/week) will be assessed using the Physical Activity and Sedentariness Questionnaire (Observatoire National de l'Activité Physique et se Sédantarité = National Observatory on Physical Activity and Sedentariness).
Muscle mass : DXA | Baseline
  Muscle mass will be measured by DXA in kg
Muscle mass : impedancemetry | Baseline
  Muscle mass will be measured by impedancemetry in kg
Bone mineral density | Baseline
  Bone mineral density will be measured by DXA in g/cm²
Resting energy metabolism | Baseline
  Resting energy metabolism will be measured by indirect calorimetry in Kcal/day

OTHER OUTCOMES:
Creation of a blood bank | Baseline
  Blood samples will be stored at the biological resource centers of Nîmes and Montpellier University Hospitals.
  As soon as the samples have been taken, the tubes are left at room temperature for about 5 minutes to coagulate (only dry tubes will coagulate). They are then centrifuged at 3800 rpm for 20 minutes at 4°C, aliquoted into cryotubes (volume 600 µl) and frozen as quickly as possible at -80°C.
Creation of a saliva bank | Baseline
  The saliva sample is taken at least 60 minutes after brushing the teeth or taking medication and at least 10 minutes after drinking (water). The subject must place the cotton swab in the mouth without touching it and leave it in the mouth for at least 3 minutes until he or she can no longer avoid swallowing the saliva produced. The subject then returns the inhibited saliva swab to the suspended container and seals the tube with the stopper. The tube was then centrifuged at 3800 rpm for 20 minutes at 4°C. The clear saliva (without residue) thus extracted is aliquoted into cryotubes (volume 600 µl) and frozen as quickly as possible at -80°C. Saliva samples will be stored at the biological resource centers of Nîmes and Montpellier University Hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Thibault MURA, Prof., Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (2):
- France (2):
  - C.H.R.U. Lapeyronie, Montpellier
  - Chu Nimes, Nîmes

IPD SHARING:
Plan to Share IPD: No
The data is managed by the BESPIM (Biostatistics, Clinical Epidemiology, Public Health and Methodological Innovation Department) at the Nîmes University Hospital. The conditions under which all or part of the research database may be transferred are decided by the research sponsor and are set out in a written contract.